CLINICAL TRIAL: NCT04733417
Title: An Exploratory Study of CDK4/6 Inhibitor SHR6390 Combined With Famitinib in the Treatment of HR + / HER2- Advanced Breast Cancer.
Brief Title: A Study of SHR6390 Combined With Famitinib in the Treatment of HR + / HER2- Advanced Breast Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-IIT-SHR6390-FMTN
Record Dates: First submitted 2020-12-30; First posted 2021-02-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-04

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — famitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR6390+famitinib (Experimental): Participants will receive SHR6390 in combination with famitinib.
  Interventions: Drug: SHR6390; Drug: famitinib

INTERVENTIONS:
Drug: SHR6390 — SHR6390 is a novel small molecule inhibitor specifically targeting the CDK4/6 pathway.
Drug: famitinib — Famitinib is a tyrosin-inhibitor agent targeting at c-Kit, VEGFR2, PDGFR, VEGFR3, Flt1 and Flt3.

SUMMARY:
The study is being conducted to assess the efficacy and safety of SHR6390 combined with famitinib in the treatment of advanced or metastatic breast cancer that progress in 1-2 line endocrine therapy.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label, Simon's two-stage design, phase II clinical trial. The purpose of this study was to evaluate the efficacy and safety of SHR6390 combined with famitinib in the treatment of HR+/HER2 advanced or metastatic breast cancer patients who have progressed during or after 1-2 line endocrine therapy. Subjects will be treated until disease progression, toxicity is intolerable, informed consent is withdrawn, and investigators determine that medication must be discontinued. Drug efficacy and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 18 to 75 years old
2. ECOG performance status 0-1;
3. Life expectancy is not less than 12 weeks;
4. Histological or cytological confirmation of HR+/HER2- recurrent/metastatic breast cancer;
5. Participants must not have received more than two prior lines of hormonal therapy;
6. Participants must not have received more than two prior lines of chemotherapy in recurrence or metastatic setting. In addition, participants must have been treated with taxanes.
7. Participants with measurable disease must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST1.1. Participants must have experienced disease recurrence or progression during or after last therapy;
8. Adequate function of major organs
9. Participants who have not received anticoagulation therapy: INR≤1.5, APTT≤1.5 ULN. Participants receiving full-dose or parenteral anticoagulation therapy had a stable dose of anticoagulant for more than 2 weeks before entering the clinical study, the result of the coagulation test is within the normal range;
10. Women of childbearing potential who have a negative pregnancy test within 14 months before enrollment and willing to use adequate contraception prior to enrollment and for the duration of study participation;
11. No radiotherapy, chemotherapy, molecular targeted therapy, immunotherapy, or surgery were received within 4 weeks before enrollment, and the toxicity of the previous treatment has been restored to ≤1 grade (such as surgery, the wound has healed completely); no endocrine therapy within 7 days before enrollment;
12. Voluntary participation in the study, signed informed consent, good compliance and willingness to cooperate with follow-up.

Exclusion Criteria:

1. Participants who previously received VEGFR TKI;
2. Participants who previously received CDK4/6 inhibitor;
3. Allergy to study drug or its components;
4. Metastasis history of the central nervous system, or brain imaging at baseline or clinical evidence suggests the presence of CNS;
5. Participated in other drug clinical trials within 4 weeks before the first dose;
6. Other malignancies within 5 years, except cured in-situ of uterine cervix carcinoma , skin basal cell carcinoma and squamous-cell carcinoma
7. History of heart disease: uncontrollable hypertension (>140/90 mm Hg), hypertensive crisis or hypertensive encephalopathy, ≥ Grade II myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (≥Grade 2, QTc interval ≥470 ms), can't stop taking drugs that may prolong QT (such as antiarrhythmic drugs) during the study; Ⅲ ~ Ⅳ stage heart failure(according to NYHA), or LVEF <50%;
8. Abnormal coagulation function (INR>1.5 or PT >ULN+4 seconds or APTT>1.5 ULN), have bleeding or thrombotic tendency or receiving thrombolytic or anticoagulant therapy;
9. A history of bleeding, with clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ≥++, or vasculitis;
10. Arterial/venous thrombosis occurred within one year before screening;
11. Tumor has invaded important blood vessels or the tumor is likely to invade important blood vessels and cause fatal hemorrhage during treatment; thyroid function is abnormal, even treatment cannot maintain normal thyroid function;
12. Urine routine test indicates urine protein ≥(++), or 24-hour urine protein ≥1.0g;
13. Long-term unhealed wounds or fractures;
14. Received major surgery or suffered severe traumatic injury, fracture or ulcer within 4 weeks after enrollment;
15. Poor absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
16. Active HBV/HCV/HIV infection;
17. Pregnant or breastfeeding women. Women of childbearing potential who have a positive pregnancy test or unwilling to use adequate contraception prior to enrollment and for the duration of study participation； Any condition which in the investigator's opinion makes the subjects unsuitable for the study participation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the proportion of patients who achieved a complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Randomization in participants with measurable disease at baseline through the end of study (12 months after the last participant is enrolled).
  Clinical benefit defined as Complete Response (CR), Partial Response (PR) or Stable Disease (SD) lasting >= 24 weeks, as determined by the Investigator according to RECIST v1.1.
Duration of Remission (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 30 months.
  Defined as the time from the first CR or PR to the first assessment of PD or death, whichever comes first.
Progression Free Survival (PFS) | Randomization to the first occurrence of disease progression as determined by the investigator according to (RECIST v1.1 ) or death from any cause, until the end of study (12 months after the last participant is enrolled)
Overall Survival (OS) | Randomization to the first occurrence of disease progression as determined by the investigator according to (RECIST v1.1 ) or death from any cause, until the end of study (12 months after the last participant is enrolled)
Safety Profile | From the first medication to 28 days after the end of treatment.
  Safety will be assessed using NCI Common Terminology Criteria for Adverse Events v5.0 (CTCAE) for reporting laboratory and non-laboratory toxicities.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Oncology, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided